CLINICAL TRIAL: NCT00565240
Title: Mid-luteal Phase Synchronization of Ovarian Folliculogenesis in Women Protocol: WHIRL-07-2971
Brief Title: Mid-luteal Phase Synchronization of Ovarian Folliculogenesis in Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Dr. Roger Pierson, University of Saskatchewan
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: WHIRL-07-59
Record Dates: First submitted 2007-11-27; First posted 2007-11-29 (Estimated); Last update posted 2010-04-22 (Estimated); Status verified 2010-04

CONDITIONS: Ovarian Follicle
Keywords: ovarian synchronization; folliculogenesis
MeSH Terms: interventions — Desogestrel; NuvaRing; Letrozole

ARMS (4):
- Oral Contraceptive (Experimental)
  Interventions: Drug: Marvelon
- Contraceptive Ring (Experimental)
  Interventions: Drug: Nuvaring
- Aromatase Inhibitors (Experimental)
  Interventions: Drug: Letrozole
- Control (No Intervention)

INTERVENTIONS:
Drug: Marvelon — oral contraceptive
  Arms: Oral Contraceptive
Drug: Nuvaring — contraceptive vaginal ring
  Arms: Contraceptive Ring
Drug: Letrozole — Aromatase Inhibitors
  Arms: Aromatase Inhibitors

SUMMARY:
We hypothesize that administration of an aromatase inhibitor (AI) and hormonal contraceptives (HC) in the mid-luteal phase of the menstrual cycle will result in atresia of the follicles in the extant wave and cause synchronous re-emergence of a new follicular wave. We anticipate that this will provide us with information to facilitate the development of a new method for ovarian synchronization; a safer, more effective ovulation induction therapy; a new method for emergency contraception; and a greater understanding of human folliculogenesis.

ELIGIBILITY:
Inclusion Criteria:

1. female volunteers of childbearing potential;
2. are first time users of OC or have discontinued OC at least 2 months prior to study entry;
3. age between 18 and 35 years old;
4. normal body mass index (18-30);
5. has signed consent form; and
6. is in good health as confirmed by medical history, physical examination

Exclusion Criteria:

1. a positive pregnancy test will automatically exclude the volunteer from participation in this study.
2. any contraindication for oral contraception use;
3. known hypersensitivity to Letrozole and co-administered medications;
4. irregular menstrual cycles;
5. ultrasonographic evidence of ovarian dysfunction, such as Polycystic Ovary Syndrome (PCOS);
6. history of pituitary tumor;
7. HIV, HBV, HCV infection;
8. vaginal infection;
9. abnormal ECG;
10. abnormal lab tests for blood profile, liver function and renal function;
11. uncontrolled diabetes and blood pressure;
12. pregnancy (suspected or diagnosed) or lactation;
13. history or suspicion of drug or alcohol abuse;
14. history of severe mental disorders;
15. participation in an investigational drug trial within the 30 days prior to selection;
16. exhibits a disorder that is a contraindication to steroid hormonal therapy, including, for example, the following conditions:

    * history of, or actual, thrombophlebitis or thromboembolic disorders.
    * history of, or actual, cerebrovascular disorders.
    * history of, or actual, myocardial infarction or coronary artery disease.
    * acute liver disease.
    * history of, or actual, benign or malignant liver tumors.
    * history of, or suspected, carcinoma of the breast.
    * known, or suspected, estrogen-dependent neoplasia.
    * undiagnosed abnormal vaginal bleeding.
    * any ocular lesion arising from ophthalmic vascular disease, such as partial or complete loss of vision or defect in visual field.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2007-11; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
To evaluate differences in the mechanisms of atresia, initiation of a new synchronous follicular wave, interval to follicle wave emergence, interval to emergence of dominant follicle, interval to menstruation, and endometrial thickness/pattern. | 24-28 days

SECONDARY OUTCOMES:
To evaluate between treatment group differences in ultrasonographic image attributes of follicular structures that develop after administration of treatment. | ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Roger A Pierson, Principal Investigator — University of Saskatchewan
Locations (1):
- Royal University Hospital, Saskatoon, Saskatchewan, Canada